CLINICAL TRIAL: NCT07325968
Title: Cardiac MRI Phenotypes and Prognostic Stratification in Myocarditis and Inflammatory Cardiomyopathy
Brief Title: Cardiac MRI in Myocarditis and Inflammatory Cardiomyopathy
Acronym: CMR-MYOINF-PRO
Status: Enrolling by invitation | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, MD, PhD, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR-MYOINF-PROG
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Myocarditis; Inflammatory Cardiomyopathy
Keywords: Cardiac MRI (CMR); Diagnosis; Prognosis; Risk stratificaiton; Radiogenomics
MeSH Terms: conditions — Myocarditis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myocarditis: Patients with myocarditis
- Inflammatory cardiomyopathy: Patients with inflammatory cardiomyopathy

SUMMARY:
Myocarditis and inflammatory cardiomyopathy represent a broad spectrum of myocardial inflammatory disorders with highly variable clinical presentations and outcomes, ranging from spontaneous recovery to progressive heart failure, malignant arrhythmias, and sudden cardiac death. Despite advances in clinical management, risk assessment in this population remains challenging due to heterogeneous disease mechanisms, dynamic disease courses, and limited tools for individualized prognostic stratification. Biopsy-proven myocarditis has been reported to be associated with a long-term mortality rate of up to 19.2% over 4.7 years.

Cardiac Magnetic Resonance Imaging (CMR) has become a central imaging modality for the evaluation of myocardial inflammation, offering comprehensive assessment of cardiac structure, function, and tissue characteristics. Beyond conventional parameters such as ventricular volumes and ejection fraction, advanced CMR techniques, including late gadolinium enhancement and parametric mapping, enable noninvasive characterization of myocardial injury, edema, and fibrosis. Emerging quantitative and distribution-based imaging markers further expand the potential of CMR to capture myocardial heterogeneity.

However, the clinical implications of diverse CMR phenotypes in myocarditis and inflammatory cardiomyopathy, particularly their value for outcome prediction and risk stratification, remain incompletely defined. This study aims to systematically evaluate CMR-derived phenotypes and their association with clinical outcomes, and to explore the role of CMR in improving risk stratification strategies in patients with myocarditis and inflammatory cardiomyopathy. Where available, genetic data will be integrated to explore potential relationships between CMR phenotypes and underlying genetic variations, further informing disease characterization and risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected acute myocarditis: clinical presentations of myocarditis, including acute chest pain, chest tightness, new-onset or worsening dyspnea, unexplained arrhythmia symptoms, and/or syncope or unexplained cardiogenic shock; diagnostic factors, including abnormal 12-lead electrocardiogram, elevated high-sensitivity cardiac troponin I level, and functional and structural abnormalities at US imaging.

Exclusion Criteria:

* Patients were excluded if they had any evidence of coronary artery disease (coronary stenosis > 50% proven by angiography) and/ or other pre-existing cardiac disease or systemic disease with interpretable symptoms, including hypertrophic cardiomyopathy, cardiac amyloidosis, arrhythmogenic right ventricular cardiomyopathy, takotsubo cardiomyopathy, ventricular noncompaction, valve disease, and pulmonary embolism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study examined patients with myocarditis or inflammatory cardiomyopathy who underwent cardiac MRI scanning.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1-10 years
  Cardiac death, heart transplantation, recurrence of myocarditis, sustained ventricular tachycardia and hospitalization for heart failure

SECONDARY OUTCOMES:
A composite of SCD and aborted SCD | 1-10 years
  SCD, defined as unexpected death within ≤1 hour of cardiac symptoms in the absence of any progressive cardiac deterioration, during sleep, or ≤24 hours of last being seen alive. Aborted SCD, defined as an appropriate implantable cardioverter defibrillator shock for ventricular arrhythmia, a nonfatal episode of ventricular fibrillation or spontaneous sustained ventricular tachycardia causing hemodynamic compromise and requiring cardioversion
Progress to dilated cardiomyopathy (DCM) | 1-10 years
  Progression to dilated cardiomyopathy will be defined by the development of left ventricular dilation accompanied by systolic dysfunction during follow-up, as assessed by cardiac imaging and clinical evaluation.